CLINICAL TRIAL: NCT00807066
Title: Multicentric Randomized Phase III Study Comparing Gefitinib Versus Platinum-Based Chemotherapy In EGFR Fish Positive NSCLC Patients (Range)
Brief Title: Randomized Gefitinib Trial
Acronym: RANGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Humanitas per la Ricerca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2008-001
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2010-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: QUALITY OF LIFE
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gefitinib
  Interventions: Drug: Gefitinib
- B (Active Comparator): Platinum based chemotherapy
  Interventions: Drug: Platinum

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250 mg/day
  Arms: A
Drug: Platinum — Platinum based chemotherapy with cycles every 21 days
  Arms: B

SUMMARY:
Patients with locally advanced (IIIB with effusion) or metastatic non-small cell lung cancer (NSCLC), EGFR FISH positive, candidate for a first-line platinum-based chemotherapy will be considered eligible for the trial. After evaluation of inclusion and exclusion criteria, and after signature of informed consent form, all eligible patients will be randomized to receive standard chemotherapy (control arm) or gefitinib (250 mg daily dose-experimental arm). Before, and in every case, no more than 4 weeks before study entry, all eligible patients will receive a complete disease staging, including thoracic and abdominal CT-scan, and blood sampling. Bronchoscopy will be done if not previously performed. Bone scan and brain CT-scan will be performed only if clinically indicated. Disease assessment will be performed every 6 weeks (every 2 cycles) for the first 6 cycles, and thereafter every 3 months, with a confirmatory evaluation in all patients with response or disease stabilization no less than 4 weeks after the response assessment, according to RECIST Criteria. A complete disease staging, including the above mentioned procedures, will be performed in case of progressive disease, and, in every cases, when patient withdrawals the trial. Following completion of protocol therapy, patients will be followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic NSCLC, EGFR FISH positive, candidate for a first-line platinum-based chemotherapy
* Histologically confirmed diagnosis of non-squamous NSCLC. Availability of tumor tissue for EGFR FISH analysis is mandatory
* Stage IIIB (with effusion) or stage IV or disease relapsed after surgery or radiotherapy and in any case not suitable for radiotherapy or surgery with curative intent
* EGFR FISH positive
* Presence of at least one measurable/evaluable not previously irradiated lesion according to RECIST criteria. Previously irradiated lesion(s) are allowed only if progressing
* ECOG performance Status 0-2
* Patient untreated with chemotherapy or EGFR targeting agents. Adjuvant chemotherapy is allowed if disease relapsed after at least 12 months after therapy completion.
* Patient candidate to standard platinum-based chemotherapy
* Patient compliance to trial procedures
* Patients must be willing to complete the FACT-L questionnaire
* Age ≥ 18 years

Exclusion Criteria:

* EGFR FISH negative tumor
* Squamous-cell carcinoma, presence of neuroendocrine features or small cell carcinoma histology
* Impossibility to ascertain EGFR FISH status
* Concomitant radiotherapy
* Less than 30 days since completion of prior wide field chest radiotherapy or persistence of any radiotherapy related toxicity.
* Symptomatic brain metastases or newly diagnosed central nervous system (CNS) metastases that have not yet been definitively treated with surgery and/or radiation. Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically stable disease and are not receiving steroid therapy.
* Known severe hypersensitivity to gefitinib or any of the excipients of this product
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* All disease sites previously included in radiotherapy fields. If all sites were included in radiotherapy fields patient is eligible only if there is evidence of progressive disease after completion of radiotherapy.
* Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uterine and squamous cell carcinoma of the skin
* Any previous chemotherapy or EGFR targeting agents
* Pregnancy or lactating. Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy
* Males must be willing to practice acceptable methods of birth control whilst taking study medication to prevent pregnancy of a partner.
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (eg, unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Concomitant use of phenytoin, carbamazepine, rifampicin, rifabutin, barbiturates or St John's Wort (Hypercium).
* Serum bilirubin greater than 3 times the upper limit of reference range (ULRR
* Alanine amino transferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases or greater than 5 times the ULRR in the presence of liver metastases.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Quality of life (FACT-L Total Score) | EVERY 3 WEEKS

SECONDARY OUTCOMES:
Time to disease progression (TTP), Objective Response Rate (ORR), overall survival (OS), and tolerability. | every two months

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Fondazione Humanitas per la Ricerca
Locations (1):
- Fondazione Humanitas per la Ricerca, Rozzano, Milan, Italy